CLINICAL TRIAL: NCT03560999
Title: Multi-Center: Non-Anesthetized Plexus Technique for Infant (BPBP) MRI Evaluation
Brief Title: Non-Anesthetized Plexus Technique for Infant (BPBP) MRI Evaluation
Acronym: NAPTIME
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Michelle James, Chief of Orthopaedic Surgery, Shriners Hospitals for Children
Other Study IDs: NCA1703
Record Dates: First submitted 2018-04-26; First posted 2018-06-19 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Brachial Plexus Palsy Due to Birth Trauma; Injury; Newborn
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators are studying the ability of a novel rapid magnetic resonance imaging (MRI) protocol to provide more accurate and earlier information about whether an infant with brachial plexus birth palsy will require nerve surgery.

DETAILED DESCRIPTION:
Brachial plexus birth palsy (BPBP) affects approximately 1 in 1,000 newborns, and though the majority of infants regain full function of the affected arm without nerve surgery, those with more severe nerve root injuries will require it. Currently, the best way to determine who will need surgery is to measure the trajectory of muscle recovery by serial clinical exams, but the optimal time for nerve surgery (before 3 months of age) is earlier than the time it usually takes to determine whether the infant needs surgery (up to 6 months.) A non-invasive diagnostic test that identifies the more severe injuries that require surgery earlier than serial exams would improve treatment timing, planning, and accuracy, and ultimately outcomes.

The investigators have developed a rapid MRI sequence with high spatial resolution and soft tissue contrast that does not require sedation or injection of a contrast agent, and that appeared to accurately assess the severity of nerve injury in infants with BPBP in a pilot study. This pilot study demonstrated that the protocol distinguishes infants who ultimately needed surgery from those who recovered spontaneously. The purpose of the current study is to enroll 100 infants at 3 centers (Shriners Hospital for Children Northern California, Boston Children's Hospital, and Gillette Children's Hospital) over a 5 year period to validate this imaging protocol as the new "gold standard" to determine whether infants with BPBP need surgery, so that individuals who need it could have surgery earlier when it is more effective, and the parents of the majority who will recover spontaneously could be spared months of worry.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of brachial plexus birth palsy.
* Age at consent ≤4 months

Exclusion Criteria:

* Bilateral brachial plexus birth palsy.
* Age at MRI <28 days or >4 months old (patients can be enrolled prior to 28 days of age, but the imaging must occur in the 28 days to 4 months' time period). The lead PI will need to approve the enrollment of a subject who will have the MRI after 90 days of age.
* Concomitant medical conditions that would preclude performance of or confound interpretation of MRI or any clinical assessment.

Ages: 0 Days to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a multicenter prospective cohort study of patients with BPBP. The study takes place at Shriners Hospitals for Children - Northern California, Boston Children's Hospital, and Gillette Children's Specialty Healthcare. All infants with BPBP between 0 and 12 weeks of age who present for treatment to a participating site will be offered participation in this study. Those infants with concomitant birth injuries that would make positioning in the MRI scanner difficult or painful (such as a birth humerus or clavicle fracture) will have their enrollment deferred. If the injury heals and the MRI can be performed within the required age range, they may be included in the study. If not, they will be excluded. Those infants who attempt to complete or actually complete the MRI scan but end up with unusable images will continue to be followed clinically, but will be removed from participation in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Whether Surgery Occurs | by 6 months of age
  The primary endpoint is the surgeon's decision for or against surgery, typically made by 6 months of age. Surgeons will make their decision based on all available clinical data, including the MRI, but will be blinded to the neuroradiologist's scoring of the SRS and its components.

SECONDARY OUTCOMES:
Intraoperative Findings | At time of surgery. Surgery occurs solely due to clinical reasons, so surgery timing (if it occurs at all) varies based on the clinical needs of the patient.
  The secondary outcome will be the surgeon's intraoperative findings during brachial plexus reconstructive microsurgery. Specifically, agreement between MRI and intraoperative findings, with respect to the level(s) and extent of injury of each nerve root and the location of root injury (pre- vs. post-ganglionic) will be determined.
AMS Scores (Hospital for Sick Children Active Movement Scale) | At follow up visits up to 30 months of age
  Active Movement Scale (AMS) measures the strength of 15 different muscles based on a scale of 0-7; 0 is no motion, and 7 is full motion against gravity.
Toronto Scores | At follow up visits up to 30 months of age
  The Toronto score also measures the strength of 15 different muscles based on a scale of 0-7; 0 is no motion, and 7 is full motion against gravity The Toronto score is a shorthand designation of the key AMS muscle strengths, in which these muscle strengths are combined (summed).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Shriners Hospitals for Children - Northern California, Sacramento, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Data will be coded and stored in a secured locked office. PHI will not be reused or disclosed to any other person or entity, except as required by law or for authorized oversight of the research project. Any disseminated data will be aggregated and coded.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT03560999/Prot_SAP_000.pdf